CLINICAL TRIAL: NCT02920294
Title: Modulation of Small Intestinal Microbial Composition and Activity,Systemic Immune Adaptation and Blood Transcriptional Changes Induced by 2-wks Consumption With 2 Fermented Milk Products;a Randomized,Exploratory,Cross-over,Double Blind,Controlled Study in Ileostomy Patients
Brief Title: Modulation of Microbial Composition in Ileostomy Patients
Acronym: INSIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: METC 163023
Record Dates: First submitted 2016-09-27; First posted 2016-09-30 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Ileostomy - Stoma
Keywords: probiotics, microbiota, ileostoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Probiotic 1 (Active Comparator): Fresh fermented dairy drink containing yoghurt ferments consumed as follows: one bottle (100g) OD for 14 consecutive days
  Interventions: Dietary Supplement: Probiotic 1
- Probiotic 2 (Active Comparator): Fresh fermented dairy drink containing probiotic strain consumed as follows: one bottle (100g) OD for 14 consecutive days
  Interventions: Dietary Supplement: Probiotic 2
- Placebo (Placebo Comparator): Acidified dairy drink without ferments consumed as follows: one bottle (100g) OD for 14 consecutive days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic 1 — Fresh fermented dairy drink containing yoghurt ferments
  Arms: Probiotic 1
Dietary Supplement: Probiotic 2 — Fresh fermented dairy drink containing probiotic strain
  Arms: Probiotic 2
Dietary Supplement: Placebo — Acidified dairy drink without ferments
  Arms: Placebo

SUMMARY:
To determine the small intestinal microbiota response in humans to dietary interventions for two consecutive weeks, and to relate this to parameters of intestinal barrier function and immune and metabolic responses in blood, as functional outcome parameters of host physiology

ELIGIBILITY:
Inclusion Criteria:

* • Ileostomy installed at least 3 years prior to participation

  * Free of any complications originating from the colectomy procedure for at least 1 yr prior to participation, with the exception of possible skin irritation at the location of the stoma
  * BMI from 18 till 28 kg/m2
  * Age from 18 till 70 years
  * Available for entire study protocol.
  * For female: If of child bearing potential, female subjects must be using or complying with methods of contraception (such as oral birth control pills, intra-uterine device, double barrier methods (like condoms and spermicide, etc.)

Exclusion Criteria:

* • History of cardiovascular, respiratory, urogenital, hepatic, haematological / immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological diseases, allergy, laboratory assessments which might limit participation in or completion of the study protocol, and/or major surgery with the exception of total colectomy, hysterectomy and/or appendectomy.

  * Subject with known lactose intolerance or with known or suspected allergy or hypersensitivity to any component of the study product(s) (milk protein for example) + sucrose + rhamnose
  * Severe gastrointestinal symptoms. In case of mild gastrointestinal symptoms, the principal investigator and the medically responsible MD will judge eligibility to participate.
  * Removal of more than 15 cm of the ileum during or at any moment after the colectomy procedure
  * Abdominal surgery interfering with gastrointestinal function, upon judgment of the principal investigator and the medically responsible MD
  * Use of medication, including proton pump inhibitors, non-steroidal anti-inflammatory drugs interfering with endpoints (but except oral contraceptives), within 14 days prior to and during participation.
  * Consumption of any probiotic or prebiotic supplements or pre- and probiotics containing food products, investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principal investigator), in the 4 weeks prior to the study and during study participation (E4 PreProbiotics).
  * Use of antibiotics in the 4 weeks prior to the start of study and during study participation
  * Prohibited use of pro-, pre- or synbiotics during study period and three months prior to start of study. A list with forbidden products will be provided'
  * History of any side effects towards intake of pro- or prebiotic supplements of any kind.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09; Primary Completion 2017-11-11 (Actual); Study Completion 2017-11-11 (Actual)

PRIMARY OUTCOMES:
Temporal microbial composition and activity in the small intestine in ileal effluent | 2 weeks intervention
  The microbiome activity will be determined as a function of the diet by double strand cDNA production and random sequencing of mRNA enriched fractions of total effluent RNA obtained from the effluent samples at the start and end of each intervention period.

SECONDARY OUTCOMES:
Small intestinal permeability by a multi sugar test (urinary recovery of test sugars) | 2 weeks intervention
Gene transcription response in blood by transcriptome patterns. | 2 weeks intervention
  Transcriptome patterns will be determined in peripheral blood mononuclear cells obtained from blood samples from the participating ileostoma patients
The levels of a panel of peripheral blood biomarkers related to immune, metabolic and hormonal status | 2 weeks intervention
  A panel of biomarkers will be determined in peripheral blood obtained at the start and end of the intervention periods
The level of whole blood immune responsiveness to a panel of standardized stimuli ex vivo | 2 weeks intervention
  Peripheral whole blood immune responsiveness towards a subset of bacterial immune-stimuli will be assessed using the standardized truculture system
Morning urine metabolome profiles | 2 weeks intervention
  The principal analytical methodology employed is mass-spectrometry profiling and can commonly provide reliable quantifications of more than 400 named-metabolites in different body-fluid samples.
Peripheral blood metabolome profiles | 2 weeks intervention
  The principal analytical methodology employed is mass-spectrometry profiling and can commonly provide reliable quantifications of more than 400 named-metabolites in different body-fluid samples.
The relative survival of bacterial strains (colony forming unit enumeration on semi-selective culture plates) | 2 weeks intervention
Short chain fatty acid profiles in ileal effluent | 2 weeks intervention
Number of participants with Gastrointestinal symptoms by Visual Analogue Scales | 2 weeks intervention
Occurrence and severity of treatment related adverse events | 2 weeks intervention

CONTACTS AND LOCATIONS:
Overall Officials: Fred Troost, PhD, Principal Investigator — Maastricht University Medical Center (MUMC+)
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zaccaria E, Klaassen T, Alleleyn AME, Boekhorst J, Smokvina T, Kleerebezem M, Troost FJ. Endogenous small intestinal microbiome determinants of transient colonisation efficiency by bacteria from fermented dairy products: a randomised controlled trial. Microbiome. 2023 Mar 7;11(1):43. doi: 10.1186/s40168-023-01491-4. PMID 36879297